CLINICAL TRIAL: NCT03400254
Title: A Phase Ib/II Trial of Gedatolisib, Hydroxychloroquine or the Combination for Prevention of Recurrent Breast Cancer ("GLACIER")
Brief Title: Gedatolisib, Hydroxychloroquine or the Combination for Prevention of Recurrent Breast Cancer ("GLACIER")
Acronym: GLACIER
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: due to business decision regarding the study drug.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Pfizer (Industry); Hoosier Cancer Research Network (Other); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UPCC 10117
Record Dates: First submitted 2018-01-11; First posted 2018-01-17 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hydroxychloroquine; gedatolisib

STUDY DESIGN:
Intervention Model Description: 24 participants in Phase Ib and 80 participants in Phase II
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase II: Arm A (Experimental): Patients will receive HCQ, 600 mg BID, for 24 weeks.
  Interventions: Drug: Hydroxychloroquine (HCQ); Drug: Gedatolisib
- Phase II: Arm B (Experimental): Patients will receive HCQ, 600 mg BID, for 24 weeks and GED x 2 weeks administered weekly, as an intravenous dose of 150 mg.
  Interventions: Drug: Hydroxychloroquine (HCQ); Drug: Gedatolisib
- Phase II: Arm C (Experimental): Patients will receive HCQ, 600 mg BID, for 24 weeks and GED x 6 weeks administered weekly, as an intravenous dose of 150 mg.
  Interventions: Drug: Hydroxychloroquine (HCQ); Drug: Gedatolisib
- Phase II: Arm D (Experimental): Patients will receive HCQ, 600 mg BID, for 24 weeks and GED x 12 weeks administered weekly, as an intravenous dose of 150 mg.
  Interventions: Drug: Hydroxychloroquine (HCQ); Drug: Gedatolisib
- Phase Ib Arm (Experimental): Patients will receive HCQ, 600 mg BID, and GED, administered weekly as an intravenous dose of 150 mg, for 6 weeks.
  Interventions: Drug: Hydroxychloroquine (HCQ); Drug: Gedatolisib

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — All patients will receive HCQ at a dose of 600 mg orally twice daily. This dose is the same in both phase Ib and phase II portions of the protocol. Capsules of HCQ are available in 200 mg strength, thus patients will initially start with 3 capsules twice daily for a total of 6 capsules per day. HCQ will be administered in divided doses (BID). When taking HCQ twice daily, the two daily doses should be taken 12 hours apart as close to 9am and 9pm as possible. Patients receiving antacids, sucralfate, cholestyramine, and/or bicarbonate should have the HCQ drug dose administered at least 1 hour before or 2 hours after these medications. Hydroxychloroquine will be obtained from the UPENN Investigational Drug Service (IDS).
Drug: Gedatolisib — Gedatolisib will be administered intravenously on a weekly dosing schedule at 150 mg IV.
  Within 3 days prior to GED dosing the patient must have an ANC >1.0 x 109/L and platelet count > 75 x 109/L. If hematologic toxicity persists, treatment should be delayed by one week and the complete blood cell count with differential and platelet count repeated. Treatment may be delayed for up to 4 consecutive weeks (28 days). If after 28 days of delay all hematologic toxicity has still not resolved to normal and non-hematologic toxicity has not resolved to <grade 1 then any further treatment with GED should be stopped.

SUMMARY:
This clinical trial will assess the safety and early efficacy of the role of gedatolisib and hydroxychloroquine in early-stage breast cancer patients with residual disease and evidence of disseminated tumor cells (DTCs) on bone marrow aspirate after neoadjuvant chemotherapy (NACT) and definitive surgery.

ELIGIBILITY:
Inclusion Criteria:

-Bone marrow aspirate after completion of neoadjuvant chemotherapy and surgery demonstrates detectable DTCs (via IHC) as performed by central laboratory assessment at Univerity of Pennsylvania.

NOTE: The criterion will be assessed AFTER confirmation of the eligibility criteria below. Patients must be pre-registered for screening of DTCs as outlined in Section 5.1 History of stage I-III histologically-confirmed primary invasive breast cancer with no evidence of recurrent local or distant disease. NOTE: Patients with bilateral breast cancer are eligible, so long as both cancers are treated with curative intent.

Any receptor status at diagnosis (by ASCO/CAP guidelines) is eligible; however, the following criteria apply:

* Patients with ER+/Her2 negative tumors must have demonstrated pathologic residual invasive disease within either the breast (with residual tumor measuring ≥ 2.5 cm) or regional lymph nodes at the time of definitive surgery following neoadjuvant therapy.
* Patients with Her2+ disease (regardless of ER status) or triple negative (ER-/PR-/Her2-) disease are eligible if there is any amount of residual disease present in the breast or regional lymph nodes at the time of definitive surgery following neoadjuvant therapy.

Prior Treatment:

* Patients must have received neoadjuvant chemotherapy prior to surgery.
* Patients must be within 24 months of undergoing definitive breast surgery post-neoadjuvant therapy. All margins of resection must be free of disease at the time of final surgical treatment.
* Patients must have completed adjuvant treatment, including post-surgery chemotherapy (if clinically indicated), radiation (if clinically indicated) and/or Her2-directed adjuvant therapy (if Her2+). Prior treatment-related toxicity must be resolved to ≤ Grade 1 with the exception of alopecia and peripheral neuropathy, prior to study enrollment..

Current/Concurrent Treatment:

* Concurrent receipt of endocrine adjuvant therapy is allowed only if therapy consists of an aromatase
* Patients will be eligible to enroll after receiving a minimum of 3 months of adjuvant endocrine therapy, to allow stabilization of side effects. Premenopausal patients on concurrent ovarian suppression are eligible. Patients on tamoxifen are ineligible due to the potential drug-drug interaction with hydroxychloroquine. Patients on any other adjuvant endocrine therapy, including any investigational therapy, are ineligible.
* Concurrent receipt of bone modifying agents (bisphosphonates or rank-ligand inhibitors) is allowed.
* No concurrent enrollment on another investigational therapy clinical trial.
* No prior therapy with a PI3Kinase inhibitor or mTOR inhibitor.
* Men and women, age ≥ 18 years.
* No contraindications to the study medications or uncontrolled medical illness.
* Adequate bone marrow, liver, and renal function and other parameters as follows:
* ANC ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Hemoglobin > 9 g/dL
* Serum bilirubin ≤ 1.5 x ULN
* ALT and AST ≤ 2.5 x ULN
* Serum creatinine ≤ 2.0 x ULN or creatinine clearance (CrCl) ≥ 30mL/min obtained within 30 days prior to registration. A calculated creatinine clearance by Cockcroft-Gault Formula is acceptable in lieu of a measured value.
* Normal coagulation studies: PT and PTT ≤ 1.5 x upper limit of normal per institutional laboratory range
* Ability to provide informed consent.
* Ability to speak and understand English

Exclusion Criteria:

* Patients with a history of another prior invasive breast cancer are ineligible. Patients with prior DCIS of the breast are eligible if this was diagnosed > 5 years prior to enrollment. Patients with prior invasive malignancy other than breast cancer are eligible if they have been disease-free for at least 5 years prior to enrollment.

Any severe and/or uncontrolled medical conditions or other conditions that could affect subject participation in the study including:

* Symptomatic congestive heart failure of New York heart Association Class III or IV
* Unstable angina pectoris, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* Severely impaired lung function with a previously documented spirometry and DLCO that is 50% of the normal predicted value (these tests not required at screening; prior results, if performed for standard of care should be referenced) and/or O2 saturation that is 88% or less at rest on room air
* Uncontrolled diabetes
* Active (acute or chronic) or uncontrolled severe infections
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis A known history of HIV seropositivity as reported by the patient. HIV testing is not required.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of hydroxychloroquine (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis. Patients receiving therapeutic anticoagulation are not eligible for study participation.

Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial and for 8 weeks after stopping study drug, by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of Gedatolisib). Inclusion of Underrepresented Populations Individuals of all races and ethnic groups are eligible for this trial. There is no bias towards age or gender.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | Approximately 4 Years
  Frequency of 'a priori' defined "severe" adverse events and any adverse event by NCI CTCAE v5 criteria (Phase Ib)
Response to Treatment | Approximately 6 Months
  "Response" to treatment is defined by a greater than or equal to 50% reduction in number of disseminated tumor cells (DTCs) at 24 weeks compared to baseline (Phase II)

SECONDARY OUTCOMES:
Occurrence of Adverse Events | Approximately 6 Months
  NCI CTCAE v5 criteria (Phase II)
Recurrence After Treatment | 3 Years
  Recurrence Free Survival (RFS)

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States